CLINICAL TRIAL: NCT06697184
Title: A Phase 1/2 Open-label Study to Investigate the Safety of Sonrotoclax Ramp-up Schedule(s) in Adult Patients With Hematological Malignancies.
Brief Title: A Study to Investigate the Safety of Novel Dose Ramp-up Schedule(s) When Initiating Sonrotoclax in Participants Treated for Blood Cancers.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-108
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lymphocytic Leukemia; CLL
Keywords: CLL previously untreated; Hematological Malignancies
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Schedule Calibration (Experimental): Participants will receive zanubrutinib monotherapy with fixed duration, followed by combination sonrotoclax with zanubrutinib at protocol-defined ramp-up schedules until target daily dose will be reached.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib
- Part 2: Schedule Expansion (Experimental): Participants will receive zanubrutinib monotherapy with fixed duration, followed by combination sonrotoclax with zanubrutinib at ramp-up schedules as determined in Part 1.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Sonrotoclax — Administered orally
  Other Names: BGB-11417
Drug: Zanubrutinib — Administered orally
  Other Names: BGB-3111

SUMMARY:
The purpose of this study is to establish the safety of novel dosing and ramp-up schedules for sonrotoclax in participants with hematological malignancies.

DETAILED DESCRIPTION:
This study will test the safety of novel sonrotoclax dosing with gradual increases of sonrotoclax dose over specified periods until the intended target daily dose is reached. The focus will be on tumor lysis syndrome (TLS) and related toxicity signals.

In the first part of the study, each ramp-up dosing schedule will first be tested in a small group of approximately 5 to 6 participants to assess safety and establish if the schedule is suitable for further testing in additional participants (schedule calibration). In the second part of the study, approved ramp-up schedules will be further assessed for safety in approximately 50 participants (schedule expansion).

Sonrotoclax is an experimental drug that works by blocking a protein called B-cell lymphoma-2 (BCL-2). This protein helps certain types of blood tumor cells to survive and grow. When sonrotoclax blocks Bcl-2 it slows down or stops the growth of tumor cells and helps them die. This can lead to improvements in patients with certain malignant diseases including Chronic Lymphocytic leukemia (CLL). The start of treatment by BCL2 inhibitor requires progressive ramp-up over the first weeks to avoid potential consequences of initial tumor cell breakage and the release of cell content in the bloodstream. Several ramp-up schedules have already been utilized so far, and this study aims to optimize the dosing schedule by evaluating novel ones as safe, while simpler and/or faster.

Zanubrutinib is a commercialized product that works by blocking a protein called Bruton's tyrosine kinase (BTK) and controlling the activity and survival of malignant B cells. Zanubrutinib has received approval in over 65 countries/regions worldwide for the treatment of adult participants with B cell malignancies, including CLL.

This study will take place at multiple centers worldwide. The overall time to participate in this study is approximately 17 months.

ELIGIBILITY:
Inclusion Criteria:

1. Stable ECOG Performance Status ≤ 2.
2. Adequate organ function and no very recent transfusion or blood growth factor
3. Participants of childbearing potential must be willing to use a highly effective method of birth control and refrain from egg donation for the duration of the study and for ≥ 90 days after the last dose of sonrotoclax or ≥ 30 days after the last dose of zanubrutinib, whichever is later.
4. Confirmed diagnosis of CLL, based on Hallek et al 2018, and requiring treatment due to certain features of their disease
5. At least 1 measurable lesion based on computed tomography (CT)/magnetic resonance imaging (MRI) and no history of prolymphocytic leukemia or Richter's transformation.

Exclusion Criteria:

1. Participants unable to comply with the requirements of the protocol
2. Serologic status reflecting active viral HBV or HCV infection
3. Positive HIV serology (HIVAb) status unless certain conditions are met.
4. Participants with any major surgical procedure ≤ 28 days before first dose of study treatment
5. Prior systemic treatment for the CLL
6. Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia requiring treatment

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience Tumor Lysis Syndrome (TLS) | Approximately 4 months
  TLS will be defined by Howard criteria during the schedule-limiting toxicity (SLT) evaluation window

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Approximately 4 months
  Safety will be assessed by monitoring and recording of all treatment emergent adverse events (AEs) graded by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 and tolerability as determined by protocol-defined Cs during the SLT evaluation window
Number of Participants with Dose Modifications During the SLT Evaluation Window | Approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (17):
- United States (6):
  - Moffitt Cancer Center, Tampa, Florida
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (6):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Genesiscare St Andrews, Adelaide, South Australia
  - Cabrini Hospital Malvern, Malvern East, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Rockingham Hospital, Cooloongup, Western Australia
  - Linear Clinical Research, Nedlands, Western Australia
- France (3):
  - Chu Dijon, Dijon
  - Chu Montpellier Hopital Saint Eloi, Montpellier
  - Iuct Oncopole, Toulouse
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - St Jamess University Hospital, Leeds

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/